CLINICAL TRIAL: NCT01216267
Title: Evaluation of Methods for the Determination of Chromogranin A in Routine Blood Samples
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Western Ontario, Canada (Other)
Responsible Party: Principal Investigator, Stanislaus H. van Uum, Principle investigator, University of Western Ontario, Canada
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HSREB16279
Record Dates: First submitted 2010-10-05; First posted 2010-10-07 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Neuroendocrine Carcinoma (Carcinoid)
Keywords: chromogranin A; neuroendocrine; carcinoid; Proton Pump Inhibitor
MeSH Terms: conditions — Carcinoma, Neuroendocrine; Carcinoid Tumor | interventions — Lansoprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- lansoprazole (Active Comparator): lansoprazole for 7 days
  Interventions: Drug: Lansoprazole

INTERVENTIONS:
Drug: Lansoprazole — lansoprazole 30 mg HS x 7 days
  Other Names: Prevacid
Drug: lansoprazole — lanzoprazole 30 mg HS for 7 days
  Other Names: pravacid

SUMMARY:
The goal of this study is to compare several methods for measurement of Chromogranin A in their ability to serve as a marker for disease activity in patients with neuroendocrine tumors.

Further, in a subgroup, we will determine if taking a proton pump inhibitor affects Chromogranin A levels.

DETAILED DESCRIPTION:
Patient group: patients with neuroendocrine tumors (active or inactive) Healthy volunteers

ELIGIBILITY:
Patients:

Inclusion Criteria:

* having neuro-endocrine disease

Exclusion Criteria:

* age below 18 or above 70 years
* prostate cancer
* kidney failure (estimated GF < 30 mL/Min)
* heart failure
* chronic atrophic gastritis
* pregnancy

Healthy subjects:

Inclusion Criteria:

* healthy

Exclusion Criteria:

* age below 18 or above 70 years
* taking any chronic medication (except OCP)
* prostate cancer
* kidney failure (estimated GFR < 30 mL/min)
* heart failure
* pheochromocytoma
* islet cell tumors
* medullary thyroid cancer
* essential hypertension
* neurofibromatosis
* use of proton pump inhibitors
* chronic atrophic gastritis
* pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2010-06; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
chromogranin A concentration serum | single time
  For determination of normal CgA range, we will recruit 60 healthy subjects (30 female, 30 male), in whom a single plasma sample will be obtained for measurement of CgA B For determination of CgA in patients with carcinoid disease (active or inactaive), we wil recruit 200 patients with carcinoid disease from our local neuroendocinre oncology clinic.

SECONDARY OUTCOMES:
Effect of PPI on chromogranin A concentration | 2 weeks
  To determine the effect of PPI on chromogranin A concentration, we will recruit a subgroup of 12 healthy subjects who will take a bedtime lansoprazole 30 mg for 7 days. Fasting serum samples for CgA will be obtained at day 7 and 1, 2, 4, and 7 days after discontinuation of the PPI.

CONTACTS AND LOCATIONS:
Overall Officials: Stan Van Uum, MD PhD, Principal Investigator — Western University, Canada
Locations (1):
- London Health Sciences Center and St. Joseph's Health Care, London, Ontario, Canada